CLINICAL TRIAL: NCT02354066
Title: The Effect of Different Foot Orthoses (Hallux Valgus Shoe; Forefoot Relief Shoe) on the Brake Response Time After Hallux Valgus and/or Additional Forefoot Surgery
Brief Title: The Effect of Foot Orthoses on the Braking Response Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dammerer Dietmar, MD, Dr. med. univ. Dietmar Dammerer, Medical University Innsbruck
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 602006052013; INS-621000-0500 (Registry Identifier: Austria: Agency for Health and Food Safety)
Record Dates: First submitted 2015-01-13; First posted 2015-02-03 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2015-09

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus surgery; forefoot surgery; brake response time; foot orthoses
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hallux valgus Surgery (Experimental): Measurement of the Brake Response Time by Pat. undergoing hallux valgus surgery (first metatarsal osteotomy, Chevron, SCARF, Austin, etc.)
  Interventions: Device: Hallux valgus Shoe; Device: Forefoot relief shoe
- Hallux valgus and forefoot surgery (Experimental): Measurement of the Brake Response Time by Pat. undergoing hallux valgus surgery (first metatarsal osteotomy; Chevron, Austin, SCARF, etc.) and additional forefoot surgery (PIP arthrodesis, second/third/etc. metatarsal osteotomy, etc.; Peg-in-Hole, WEIL-Osteotomy, etc.)
  Interventions: Device: Hallux valgus Shoe; Device: Forefoot relief shoe
- Control Run (Experimental): Measurement of the Brake Response Time by Healthy Participants; control run; brake response time measurement with normal shoe and both foot orthoses
  Interventions: Device: Hallux valgus Shoe; Device: Forefoot relief shoe; Device: Retail Shoe

INTERVENTIONS:
Device: Hallux valgus Shoe — Brake response measurement after surgery with this foot orthosis
  Other Names: ofa® hallux valgus shoe
Device: Forefoot relief shoe — Brake response measurement after surgery with this foot orthosis
  Other Names: GloboPed® Forefoot relief orthosis
Device: Retail Shoe — Brake response time measurement before surgery (control run)
  Arms: Control Run

SUMMARY:
Patients often seek advice from their treating doctor if they are able to drive with a foot orthosis after a first metatarsal osteotomy for symptomatic hallux valgus and/or after an additional forefoot surgery. This challenging question is of obvious importance for the patient and other road users. Previous studies already issued driving ability after different orthopedic procedures and with knee and ankle devices on the brake reaction time but missed to address the same for foot orthoses after hallux valgus or forefoot surgery.

This missing evidence made us evaluate the influence of wearing a foot orthosis after a first metatarsal osteotomy or forefoot surgery on driving ability (brake response time; BRT).

The overall time frame is about nine weeks; each appointment for BRT measurement takes about fifteen to twenty minutes. The first BRT measurement is one day before the foot surgery without a foot orthosis (normal shoe)and with the orthoses (control run) (1) at two days (2), two weeks (3), four weeks (4) and six weeks (5) after the operation with a HVS and a FRS and eight weeks postoperative without a foot orthoses (6).

DETAILED DESCRIPTION:
The purpose of this study is to asses driving ability (brake response time) and the influence of two types of different foot orthoses after foot surgery.

Therefore we have two groups:

1. Hallux valgus surgery (Chevron, Austin, SCARF, Akin etc.)
2. Hallux valgus and additional forefoot surgery (Chevron, Austin, SCARF, Akin etc. and WEIL - Osteotomy, Peg-in-Hole, etc.)

BRT (brake response time) is assessed with commonly used right-sided hallux valgus shoes (HVS) and forefoot relief shoes (FRS). We measure the BRT at six different time points: one day before surgery without a foot orthosis (normal shoe)and with the orthoses (control run) (1) at two days (2), two weeks (3), four weeks (4) and six weeks (5) after the operation with a HVS and a FRS and eight weeks postoperative without a foot orthoses (6). The overall time frame is about nine weeks; each appointment for BRT measurement takes about fifteen to twenty minutes.

The BRT was assessed using a custom-made driving simulator as used in previously published studies. Participants were instructed to apply the brake pedal exclusively with the right foot as quickly as possible on a visual stimulus. The time interval until the subject operated the brake was measured 20 times, averaged and then taken as BRT value.

ELIGIBILITY:
Inclusion Criteria:

* participants must have a valid driver´s license,
* used the right foot exclusively for accelerating and braking,
* free of any medical condition that could impair the ability to drive

Exclusion Criteria:

* taking medications that could affect reaction time (e.g. benzodiazepines and over-the-counter allergy and cold medications)
* had a history of alcohol or drug abuse,
* a central nervous system disorder such as epilepsy,
* a metabolic disorder,
* a psychiatric disorder,
* musculoskeletal disease,
* any visual acuity disorder (macular degeneration etc.; glasses allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Brake response time after hallux valgus surgery with the investigated foot orthoses | July 2015 (The overall time frame is about nine weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Biedermann, Priv.Doz.Dr., Principal Investigator — University Hospital of Innsbruck, Anichstraße 35, 6020 Innsbruck, Austria, Europe
Locations (1):
- Department of Orthopedic; Medical University of Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Dammerer D, Giesinger JM, Biedermann R, Haid C, Krismer M, Liebensteiner M. Effect of knee brace type on braking response time during automobile driving. Arthroscopy. 2015 Mar;31(3):404-9. doi: 10.1016/j.arthro.2014.09.003. Epub 2014 Nov 8. PMID 25442646
- [Background] Liebensteiner MC, Rochau H, Renz P, Smekal V, Rosenberger R, Birkfellner F, Haid C, Krismer M. Brake response time returns to the pre-surgical level 6 weeks after unicompartmental knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1926-31. doi: 10.1007/s00167-014-3050-1. Epub 2014 May 15. PMID 24832693
- [Derived] Dammerer D, Braito M, Biedermann R, Ban M, Giesinger J, Haid C, Liebensteiner MC, Kaufmann G. Effect of surgical shoes on brake response time after first metatarsal osteotomy--a prospective cohort study. J Orthop Surg Res. 2016 Jan 20;11:14. doi: 10.1186/s13018-016-0350-9. PMID 26792613